CLINICAL TRIAL: NCT00315003
Title: Multinational, Randomized, Double-Blind, Double-Dummy, Comparative Study to Evaluate the Efficacy and Safety of 5 Days Telithromycin 25mg/kg od Versus 5 Days Azithromycin 10 mg/kg od Followed by 5 mg/kg od for 4 Days, in Children With Acute Otitis Media
Brief Title: TELI COM - Telithromycin in Children With Otitis Media
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Pediatric development program terminated by sponsor
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6132; HMR3647B/3002
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Otitis Media, Suppurative; Otitis Media, Purulent
Keywords: Otitis Media; Suppurative; Purulent; Ketolide; Azithromycin; Telithromycin; Controlled Clinical Trials
MeSH Terms: conditions — Otitis Media, Suppurative; Otitis Media; Suppuration | interventions — telithromycin; Azithromycin

INTERVENTIONS:
Drug: Telithromycin
Drug: Azithromycin

SUMMARY:
This is a multinational, randomized (1:1), double-blind, double-dummy, comparative, 2- treatmentgroup study in children (age range: ≥6 months and <72 months [< 6 years of age]) with AOM.Subjects will be randomized to receive either telithromycin (50 mg/mL) oral suspension 25 mg/kgonce daily for 5 days or azithromycin (40 mg/mL) oral suspension (10 mg/kg once on Day 1, followed by 5 mg/kg once daily on Days 2-5, not to exceed 500 mg onDay 1 and 250 mg/day from Days 2 - 5. Matching placebo suspensions for telithromycin and azithromycin will also be dispensed to provide blinding for the different treatment regimens.Assessments and reporting of safety will be carried out at all visits.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria will be considered for enrollment into the study:

* Subjects ≥6 months and <72 months (< 6 years) of age;
* Recent (within the last 72 hours) and rapid onset of AOM symptoms and signs;
* The presence of MEF on otoscopy indicated by a bulging tympanic membrane;
* Otalgia or ear tugging or touching within the last 24 hours that interferes with or precludes normal activity or sleep;
* At least 1 of the following clinical findings not specific to AOM: fever, vomiting, diarrhea, anorexia, sleep disturbance, or irritability;
* Caregiver-reported AOM symptoms sufficient for entry according to protocol criteria.
* Caregiver-reported AOM symptoms diary
* Tympanometry exhibiting:

  * Type B curve or positive pressure peak curves.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

* Uncertain diagnosis of AOM or mild to moderate symptoms and signs of AOM that would make the subject a candidate for observation and analgesic therapy with observation for 2-3 days.
* Otorrhea or tympanostomy tube present in the ear to be evaluated;
* Otitis externa;
* Down syndrome, cleft palate, craniofacial disorders, cystic fibrosis/mucoviscidosis, immotile cilia syndrome, congenital immunodeficiency or acquired immunodeficiency syndrome with <25% CD4 count or requiring prophylaxis for Pneumocystis jiroveci (carinii) or requiring treatment for an opportunistic infection;
* Known congenital long QT syndrome;
* Known or suspected uncorrected hypokalemia (≤3 mmol/L [mEq/L]), hypomagnesemia, bradycardia (<50 bpm);
* Myasthenia gravis;
* Known impaired renal function, as shown by creatinine clearance ≤25 mL/min;
* History of hypersensitivity or intolerance to macrolides or azithromycin;
* Previous enrollment in this study or previous treatment with telithromycin;
* Children of the investigator or subinvestigator, research assistant, pharmacist, study coordinator, other staff, or relative thereof directly involved in the conduct of the protocol.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1500
Dates: Start 2006-01; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variables will be time to symptom resolution (TSR) and clinical cure at theposttherapy/TOC Visit 3.

SECONDARY OUTCOMES:
Adverse events (AEs) reported by subjects, their parents/legally authorized representative, orobserved by the investigators will be recorded throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (13):
- Sanofi-Aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis, Buenos Aires, Argentina
- Sanofi-Aventis, São Paulo, Brazil
- Sanofi-Aventis, Laval, Canada
- Sanofi-Aventis, Providencia, Santiago Metropolitan, Chile
- Sanofi-Aventis, Bogotá, Colombia
- Sanofi-Aventis, San José, Costa Rica
- Sanofi-Aventis, Prague, Czechia
- Sanofi-Aventis, Santo Domingo, Dominican Republic
- Sanofi-Aventis, Guatemala City, Guatemala
- Sanofi-Aventis, Israel, Israel
- Sanofi-Aventis, Panama City, Panama
- Sanofi-Aventis, Lima, Peru